CLINICAL TRIAL: NCT00608816
Title: Hypoglycemia Associated Autonomic Failure in Type 1 DM, Question 4
Brief Title: Hypoglycemia Associated Autonomic Failure in Type 1 DM, Q4
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Steve Davis, Chairman of Medicine, University of Maryland, Baltimore, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: IRB #040910-HAAF in T1DM, Q4; Ro1 DK06903-03
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Type 1 Diabetes
Keywords: epinephrine
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Hyperinsulinemic euglycemic glucose clamp study on day 1 Hyperinsulinemic euglycemic clamp study on day 2 with epinephrine infusion
  Interventions: Drug: epinephrine
- 2 (Experimental): Hyperinsulinemic hypoglycemic glucose clamp x 2 on day 1 Hyperinsulinemic euglycemic clamp with epinephrine infusion on Day 2
  Interventions: Drug: epinephrine

INTERVENTIONS:
Drug: epinephrine — Epinephrine 0.06 µg/kg/min infusion during a two hour experimental period on Day 2
  Arms: 1
Drug: epinephrine — Epinephrine 0.06 µg/kg/min infusion during two hour experimental period on Day 2
  Arms: 2

SUMMARY:
Epinephrine is one of the important hormones in the defense of hypoglycemia. We will test the hypothesis that antecedent hypoglycemia will blunt the metabolic, neuroendocrine and cardiovascular effects of subsequent epinephrine infusion in Type 1 DM.

DETAILED DESCRIPTION:
When a person had previously experienced bouts of low blood sugar, or hypoglycemia, his or her counterregulatory responses to hypoglycemia would be weakened. This is especially true and important for a person with Type 1 diabetes, because it will cause him or her to be vulnerable to another bout of hypoglycemia, and cause hypoglycemia unawareness, which can lead to serious or even life-threatening consequences. Epinephrine is one of the important hormones in the defense of hypoglycemia. We will test the hypothesis that antecedent hypoglycemia will blunt the metabolic, neuroendocrine and cardiovascular effects of subsequent epinephrine infusion in Type 1 DM.

ELIGIBILITY:
Inclusion Criteria:

* 28 (14 males, 14 females) conventionally treated Type 1 diabetic patients with HA1C > 8.5%
* 28 (14 males, 14 females) intensively treated Type 1 diabetic patients with HA1C < 7%
* 28 (14 males, 14 females) non-diabetic controls
* Age 18-45 yr.
* Had diabetes for 2-15 years if diabetic subject
* No clinical evidence of diabetic tissue complications, no cardiovascular disease
* Body mass index 21-27kg · m-2
* Normal bedside autonomic function
* Normal results of routine blood test to screen for hepatic, renal, and hematological abnormalities
* Female volunteers of childbearing potential: negative HCG pregnancy test

Exclusion Criteria:

* Prior history of poor health: any current or prior disease condition that alters carbohydrate metabolism and prior cardiac events and/or evidence for cardiac disease
* Hemoglobin of less than 12 g/dl
* Abnormal results following screening tests
* Pregnancy
* Subjects unable to give voluntary informed consent
* Subjects with a recent medical illness
* Subjects with known liver or kidney disease
* Subjects taking steroids
* Subjects taking beta blockers
* Subjects on anticoagulant drugs, anemic, or with known bleeding diseases

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
catecholamine levels | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, Principal Investigator — Vanderbilt University